CLINICAL TRIAL: NCT04570579
Title: Impact of a Novel Extended Depth of Focus Intraocular Lens on Visual and Lifestyle Enhancement
Status: Active, not recruiting | Type: Observational
Sponsor: Alanna Nattis, DO (Other)
Responsible Party: Sponsor-Investigator, Alanna Nattis, DO, Director of Clinical Research, Ophthalmologist, Sight Medical Doctors PLLC
Organization: Sight Medical Doctors PLLC (Other)
Other Study IDs: EDOF Lifestyle Enhancement
Record Dates: First submitted 2020-09-13; First posted 2020-09-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cataract; Cataract Senile; Presbyopia
Keywords: cataract; presbyopia-correcting intraocular lens; cataract surgery; refractive cataract surgery
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational cohort: This is a prospective, nonrandomized study of patients undergoing bilateral cataract surgery with implantation of the spherical Vivity and/or Vivity toric IOL. Preoperative patient data such as age, sex, prior ocular history, medical history, and intraocular lens calculations/formulae used will be recorded. Uncorrected and best-corrected visual acuity will be measured at distance (4m), intermediate (60cm) and near (40cm). All 3 surveys will be administered prior to surgery (at baseline) and at 3 months postoperative, regarding spectacle independence, visual disturbances, and visual quality. A proper perioperative record will be maintained, documenting planned IOL implantation, actual IOL implant used, use of femtosecond laser, use of intraoperative aberrometry, and use of pupillary expansion devices. Patients will be examined 1 day ("postoperative day 1)", 1 week ("postoperative week 1"), 1 month ("postoperative month 1") and 3 months ("postoperative month 3") following surgery.
  Interventions: Device: Vivity Extended Depth of Focus Intraocular Lens

INTERVENTIONS:
Device: Vivity Extended Depth of Focus Intraocular Lens — Patients selected to have bilateral sequential cataract surgery using the Vivity (spherical and/or toric where applicable) intraocular lens implant will subsequently be offered enrollment into this observational study. Visual outcomes will be recorded at postoperative day 1, week 1, month 1 and month 3.

SUMMARY:
The introduction of presbyopia-correcting intraocular lenses (PC-IOLs) has provided cataract and refractive surgeons the ability to provide patients with a wider range of visual success and spectacle independence post-cataract surgery.Multifocal (MFIOL) IOLs have the ability to provide near and distance vision, and in the case of trifocal IOLs, near, intermediate and distance. Despite the significant technological evolution of MFIOL's, the potential for visual disturbances, such as glare, halos and starbursts still exists-and in much greater frequency compared to their monofocal counterparts.

Extended depth of focus (EDOF) IOLs aim to provide patients with a functional range of vision, with a similar visual disturbance profile to a monofocal lens. In this way, this subset of PC-IOL's can offer patients some degree of spectacle independence, with a significantly lower incidence of visual disturbances.

The Vivity Extended Vision IOL is the first of its kind to offer Wavefront Stretching technology, providing patients with an excellent extended range of vision from intermediate to distance, as well as some functional near vision. Prior studies have demonstrated very good vision in both bright and dim lighting conditions, as well as a high degree of spectacle independence with the Vivity IOL, as compared to a monofocal IOL.

Studies evaluating the ability of the Vivity IOL to provide a significant impact on patient lifestyle (e.g. patient independence from spectacles for most activities with a low rate of visual disturbances) in the United States in a 'real-world' setting have yet to be performed. In addition, influence of pre-and-perioperative variables such as sex, age, prior refractive surgery, IOL formula used, axial length, astigmatism, use of intraoperative aberrometry, femtosecond laser and pupillary expansion devices has yet to be evaluated on the postoperative success of this IOL.

This study will be comprised of patients with visually significant cataracts who will undergo cataract extraction with implantation of the spherical and/or toric models of the Vivity Extended Vision (Alcon, Fort Worth TX) intraocular lens. Upon decision of the patient and surgeon to undergo surgery, patients will be offered the option to enroll in this observational study.

DETAILED DESCRIPTION:
Presbyopia-correcting intraocular lenses (PC-IOLs) provide cataract and refractive surgeons with an effective treatment option for presbyopia, allowing patients increased spectacle independence post-cataract surgery. Different IOL designs have been developed based on differing optical principals, such as diffractive, refractive and extended depth of focus (EDOF) design. Most commercially available MFIOLs have two optical zones, one that provides distance vision, and the second that provides near vision (i.e. "bifocal IOLs"). Most recently, trifocal IOLs have been released, with the aim of providing a third (intermediate) focal point, and hence an extended range of vision in pseudophakic patients. While being able to provide patients with near, intermediate and distance vision, most MFIOL's carry the risk of increased visual disturbances, such as glare, starbursts, and halos, which for a small percentage of patients may become quite bothersome or even debilitating.

Extended depth of focus (EDOF) IOLs aim to provide an extended range of vision from intermediate to distance, with a similar visual disturbance profile to their monofocal counterparts. Prior to recent FDA approval, there was only one other EDOF IOL on the market in the US, which, although provides an extended visual range, still had a significant incidence of starbursts and visual disturbances in some patients. FDA approved in February 2020, the Vivity Extended Vision Lens has demonstrated the ability to provide patients with an extended range of vision, excellent contrast sensitivity and visual disturbance profile comparable to a monofocal IOL, as well as high rates of spectacle independence for most activities.

The Vivity Extended Vision IOL (Alcon Laboratories, Fort Worth TX) is an EDOF IOL made of hydrophobic acrylic. This non-diffractive lens was designed to mitigate the effect of presbyopia by providing an extended depth of focus through patented Wavefront Shaping technology. In clinical trials, Vivity has demonstrated significantly better intermediate and near vision as compared to a monofocal IOL, as well as superior spectacle independence scores. Additionally, a validated questionnaire regarding visual disturbances showed the Vivity to have comparable rates of starburst, glare and halos to its monofocal counterpart.

In an era where intermediate vision has become very important (e.g. using laptops, tablets, seeing the dashboard in a car), many patients express desire for visual correction at all possible focal points. Vivity appears to deliver this with minimal visual side effects-even less so as compared to other MFIOL's. This is a valuable aspect of Vivity; spectacle independence is an important factor for many patients-however if this is coupled with debilitating glare, haloes or other visual disturbances, dissatisfaction will ultimately result.

Multiple studies have explored variables that may influence postoperative success of these MFIOLs, including the impact of dry eye, prior corneal refractive surgery, and proper preoperative consent/expectations.

A study has yet to be performed evaluating not only preoperative factors, such as astigmatism, and prior corneal refractive surgery, but also perioperative and intraoperative factors that may also play a role in success of the Vivity IOL implant. In this prospective, nonrandomized "real-world" study, the impact of perioperative factors, such as IOL formulae used, use of femtosecond laser, use of intraoperative aberrometry, as well use of pupillary expansion devices on surgical success will be evaluated. Surgical success will be defined as uncorrected distance, intermediate and near visual acuity (UDVA, UIVA and UNVA, respectively) of 20/40 or better (both monocular and binocular) as well as high levels of patient satisfaction, which will be recorded with a Visual Disturbance Questionnaire, Spectacle Independence Questionnaire, and Visual Quality Questionnaire.

Results will provide never-before-published data on important preoperative as well as perioperative factors that may influence success and patient satisfaction with Vivity IOL implantation

ELIGIBILITY:
Inclusion Criteria:

* Visually significant bilateral cataracts, with planned cataract extraction using phacoemulsification and clear corneal incision
* Ability to comprehend and willing to sign informed consent
* Ability to complete all required postoperative follow up procedures.
* 18 years or older
* male or female

Exclusion Criteria:

* Patients who lack ability to consent, and who cannot provide clear understanding of the surgical procedure as well as possible adverse side effects (e.g. dysphotopsias) of the IOL will be excluded
* Patients who are professional night drivers, pilots and those with other occupations for whom induced dysphotopsia could put their career at risk will be excluded
* Patients who have preexisting significant ocular pathology, including severe dry eye, retina, optic nerve (including moderate-severe glaucoma) and corneal pathologies (e.g. corneal dystrophy, edema, significant scarring), limiting or affecting visual potential, in the opinion of the surgeon, will be excluded
* Patients whose IOL calculations are outside the range available for the Vivity IOL will be excluded.
* Patients who have history of past eye trauma with evidence of/suspected zonular laxity, and those with pseudoexfoliation will be excluded.
* Patients with prior corneal surgery (namely, radial keratotomy (RK), corneal transplantation of any kind) will be excluded from the study (post-myopic and hyperopic LASIK and PRK patients will be permitted to participate in the study).
* Pregnant and/or lactating patients will be excluded from the study.
* Patients with perioperative or intraoperative complications that do not allow for implantation of the Vivity IOL will be excluded.
* Inability to implant the Vivity IOL will cause immediate release from the study with documented rationale for exit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from a large clinical ophthalmic practice after having been determined to have visually significant cataracts requiring cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual success - uncorrected distance visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in uncorrected distance visual acuity between baseline and at 3 months postoperative will be assessed.
Visual success- uncorrected intermediate visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in uncorrected intermediate visual acuity between baseline and at 3 months postoperative will be assessed.
Visual success- uncorrected near visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in uncorrected near visual acuity between baseline and at 3 months postoperative will be assessed.
Visual success - best corrected distance visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in best-corrected distance visual acuity between baseline and at 3 months postoperative will be assessed.
Visual success- best-corrected intermediate visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in best-corrected intermediate visual acuity between baseline and at 3 months postoperative will be assessed.
Visual success- best-corrected near visual acuity | Change in visual acuity outcomes will be assessed at baseline and compared to postoperative month 3
  Change in best-corrected near visual acuity between baseline and at 3 months postoperative will be assessed.
Visual quality of life measures - visual disturbances | Questionnaires will be administered at baseline visit (preoperative) and at 3 months postoperative
  Change in responses in regard to patient lifestyle satisfaction using a Visual Disturbance Questionnaire at baseline and 3 months postoperative will be assessed. This will be assessed on a scale of 0 - 4 in severity (0 = no disturbance, 4 = very bothersome disturbance). Total scores will be tallied and compared between baseline and postoperative month 3 responses.
Visual quality of life measures - Visual quality | Questionnaires will be administered at baseline visit (preoperative) and at 3 months postoperative
  Change in responses in regard to patient lifestyle satisfaction using a Visual Quality Questionnaire at baseline and 3 months postoperative will be assessed. This will be assessed on a scale of 1 - 5 in severity (1 = no issues with vision interfering with daily activities, 5 = vision interfering with nearly every activity listed). Total scores will be tallied and compared between baseline and postoperative month 3 responses.
Visual quality of life measures - spectacle independence | Questionnaires will be administered at baseline visit (preoperative) and at 3 months postoperative
  Change in responses in regard to patient lifestyle satisfaction using a Spectacle Independence Questionnaire at baseline and 3 months postoperative will be assessed. This will be assessed on a scale of 0 - 4 in severity (0 = never using spectacles for activities, 4 = always using spectacles for every activity listed). Total scores will be tallied and compared between baseline and postoperative month 3 responses.

OTHER OUTCOMES:
Adverse events | Safety measures and assessment for adverse events will be assessed at all time points (baseline, postoperative day 1, postoperative week 1, postoperative month 1, postoperative month 3)
  Adverse events (e.g. surgical complications) in relation to Vivity IOL implantation will be evaluated at each time point. Any adverse events will be documented/reported and treated, if necessary

CONTACTS AND LOCATIONS:
Locations (1):
- SightMD, Babylon, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to make IPD data available to other researchers.

REFERENCES:
- [Background] Lichtinger A, Rootman DS. Intraocular lenses for presbyopia correction: past, present, and future. Curr Opin Ophthalmol. 2012 Jan;23(1):40-6. doi: 10.1097/ICU.0b013e32834cd5be. PMID 22081027
- [Background] Alfonso JF, Fernandez-Vega L, Puchades C, Montes-Mico R. Intermediate visual function with different multifocal intraocular lens models. J Cataract Refract Surg. 2010 May;36(5):733-9. doi: 10.1016/j.jcrs.2009.11.018. PMID 20457363
- [Background] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Background] Wang SY, Stem MS, Oren G, Shtein R, Lichter PR. Patient-centered and visual quality outcomes of premium cataract surgery: a systematic review. Eur J Ophthalmol. 2017 Jun 26;27(4):387-401. doi: 10.5301/ejo.5000978. Epub 2017 Apr 24. PMID 28574135
- [Background] Cochener B, Boutillier G, Lamard M, Auberger-Zagnoli C. A Comparative Evaluation of a New Generation of Diffractive Trifocal and Extended Depth of Focus Intraocular Lenses. J Refract Surg. 2018 Aug 1;34(8):507-514. doi: 10.3928/1081597X-20180530-02. PMID 30089179
- [Background] de Medeiros AL, Jones Saraiva F, Iguma CI, Kniggendorf DV, Alves G, Chaves MAPD, Vilar C, Motta AFP, Carricondo PC, Takashi Nakano C, Nose W, Hida WT. Comparison of visual outcomes after bilateral implantation of two intraocular lenses with distinct diffractive optics. Clin Ophthalmol. 2019 Aug 29;13:1657-1663. doi: 10.2147/OPTH.S202895. eCollection 2019. PMID 31695317
- [Background] Savini G, Schiano-Lomoriello D, Balducci N, Barboni P. Visual Performance of a New Extended Depth-of-Focus Intraocular Lens Compared to a Distance-Dominant Diffractive Multifocal Intraocular Lens. J Refract Surg. 2018 Apr 1;34(4):228-235. doi: 10.3928/1081597X-20180125-01. PMID 29634837
- [Background] Williams D, Yoon GY, Porter J, Guirao A, Hofer H, Cox I. Visual benefit of correcting higher order aberrations of the eye. J Refract Surg. 2000 Sep-Oct;16(5):S554-9. doi: 10.3928/1081-597X-20000901-12. PMID 11019871
- See also: FDA Summary of Safety and Effectiveness Data: Vivity Extended Vision IOL — https://www.accessdata.fda.gov/cdrh_docs/pdf/P930014S126B.pdf
- See also: Acrysof IQ Vivity Intraocular Lens Product Information — https://www.accessdata.fda.gov/cdrh_docs/pdf/P930014S126C.pdf